CLINICAL TRIAL: NCT00909272
Title: Ultrasound Guided Diagnostic Lumbar Medial Branch Blocks
Status: Withdrawn | Type: Observational
Why Stopped: One of the investigators has left the institution
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Other Study IDs: 09-039-D
Record Dates: First submitted 2009-05-22; First posted 2009-05-27 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Back Pain
Keywords: ultrasound; diagnostic; lumbar; median branch; block; Lumbar facet joint pain
MeSH Terms: conditions — Back Pain; Disease; Bites and Stings

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- US-guided lumbar medial branch block: Patients who have low back pain and/or leg pain due to possible lumbar facet joint disease .
  Interventions: Procedure: Lumbar medial branch block
- Cadavers for Ultrasound landmarks: Cadavers donated to the Department of Anatomy in McMaster University will be used to determine the landmarks for ultrasound.
  Interventions: Procedure: Ultrasound landmarks

INTERVENTIONS:
Procedure: Lumbar medial branch block — The ultrasound probe will be placed perpendicular to skin along the midline of lumbar spinous process on longitudinal view first to count the lumbar level. The midpoint of each lumbar level will be marked on the longitudinal view and then will be rotated ninety degrees counter clockwise to axial view to locate the facet joint and the transverse process of lumbar spine. A #22 gauge 10cm long Quincke spinal needle will be inserted to the target area using in plane approach on the axial view. Then the probe will be rotated ninety degrees clockwise to longitudinal view to ensure needle tip is placed on the cephalad aspect of the transverse process. It will then be immediately confirmed by C-arm fluoroscopy on oblique view.
  Groups: US-guided lumbar medial branch block
Procedure: Ultrasound landmarks — The target point is the superior medial aspect of transverse process of lumbar spine from L3 to S1. A #22 gauge 10cm long Quincke spinal needle will be use for needle placement. Needle placement will be visualized with ultrasound. Practice on cadavers with 3 different operators and see if results are reproducible. Verify with fluoroscopy.
  Groups: Cadavers for Ultrasound landmarks

SUMMARY:
Can an ultrasound machine be used to perform a diagnostic lumbar medial branch block?

DETAILED DESCRIPTION:
The diagnostic lumbar medial branch block for low back and radiating to lower extremity due to lumbar facet joint pain has been traditionally done under fluoroscopic guidance. Some recent studies have shown that the diagnostic lumbar medial branch may alternatively be done under ultrasound guidance. This proposed technique has many advantages, avoid radiation exposure and decrease waiting period for patients to have a pain procedure for low back pain. The time taken, patients' satisfaction score, pain score, the distance the needle tip placed under ultrasound and the ideal position visualized under fluoroscopy will be measured. This study will be done in 2 parts. The first part will determine landmarks for ultrasound. It will involve using 5 cadavers. The second part of the study will involve 25 patients. The needles will be placed initially with ultrasound and then will be verified with C-arm fluoroscopy. Certain criteria will be used to determine its feasibility, for example, less than 20 minutes, less than 5 mm.

ELIGIBILITY:
Inclusion Criteria:

* Low back and/or leg pain due to possible lumbar facet joint disease

Exclusion Criteria:

* patient with BMI>35
* coagulopathy
* allergy to local anesthetic and ultrasound gel
* patient unable to fill out post procedure pain diary

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care pain clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Perform a diagnostic lumbar medial branch block using ultrasound guidance, decide if it's practical to perform it, whether patients can tolerate it, can it be performed in a timely manner and the # of needle adjustments required to get target points. | At time of procedure

SECONDARY OUTCOMES:
Does this procedure correlate with other known procedures, by the distance between the needle tip placed under the ultrasound and the superior medial aspect of transverse process of lumbar spine L3 to S1 visualized under C-arm fluoroscopy. | At time of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Park, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences-General Location, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Shim JK, Moon JC, Yoon KB, Kim WO, Yoon DM. Ultrasound-guided lumbar medial-branch block: a clinical study with fluoroscopy control. Reg Anesth Pain Med. 2006 Sep-Oct;31(5):451-4. doi: 10.1016/j.rapm.2006.06.246. PMID 16952818